CLINICAL TRIAL: NCT07297849
Title: The Effect of Eyelid Closure on the Quality Index of Keratometric Measurements: a Non-controlled Interventional Study
Brief Title: Eyelid Closure in Keratometry
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Head of Department, Vienna Institute for Research in Ocular Surgery
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: EK 24-111-0824
Record Dates: First submitted 2025-12-02; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Dry Eye; Ocular Surface Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with a keratometrical warning index (Experimental): The following measurements will be performed in the mentioned order during the visit 1 only in the randomized study eye:
  1. First and second biometry using IOLMaster® 700 (2x, 3 minutes pause between the measurements, eyes open, normal blinking)
  2. Eyelid closure for 3 minutes
  3. Third biometry using IOLMaster® 700 (1x) right after opening of the eyelid
  4. Eyelid closure for 3 minutes
  5. Fourth biometry using IOLMaster® 700 (1x) right after opening of the eyelid
  Interventions: Behavioral: Eyelid closure for 3 minutes

INTERVENTIONS:
Behavioral: Eyelid closure for 3 minutes — Patients will be advised to close their eyes for 3 minutes before the third and before the fourth study measurement.

SUMMARY:
Cataract surgery is one of the most common performed surgeries in the world. While in the early beginnings of cataract surgery, visual rehabilitation was the main goal of the procedure, refractive outcome and subsequent relative spectacles independency is gaining increasing importance in patients' demands. Due to the improvements in measurement techniques and prediction formulas, the prediction of postoperative refraction is possible with high accuracy. However, there are still some sources of error that lead to deviations of predicted postoperative refraction. For instance, it was shown that tear film osmolarity, an established biomarker for dry eye disease (DED), plays an important role in preoperative precision of keratometry measurements. Keratometry, the measurement of corneal curvature, is an important part of preoperative biometry. Errors in preoperative keratometry measurements lead to nearly one-to-one deviations from the predicted refraction. Therefore, proper keratometry measurements are a key element in intraocular lens (IOL) power calculations. To counteract the issue of DED in preoperative biometry, the principle of using lubricating eye drops before ocular biometry has been investigated and it was shown that the use of ocular lubricants may lead to increased variability of keratometry measurements. From our clinical observations, another possible mechanism to improve keratometry is eyelid closure for some minutes. In contrast to the long-term use of ocular lubricants to stabilize the tear film, eyelid closure is an easy and fast intervention to possibly improve the precision of keratometry measurements. Additionally, a clinical trial investigating the usage of lubricating eye drops for two weeks found no improvement of variability of keratometry in DED patients.

Therefore, this study aims to investigate the effect of eyelid closure on the quality index of keratometric measurements in patients with a warning for the quality of keratometric measurements. For this purpose, a single study day including 4 repeated measurements (2 without and 2 with lid closure for 3 minutes) using an ocular biometer (IOLMaster700) will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Written informed consent
* Keratometry quality index "warning"

Exclusion Criteria:

* Severe corneal conditions that may compromise corneal integrity (such as corneal scarring, etc.)
* Pregnancy (pregnancy test will be taken in women of reproductive age), nursing women
* Ocular surgery in the study eye in the three months preceding the study
* Inability of visual fixation (e.g. in patients with nystagmus)
* Inability of eyelid closure (e.g. in patients with facial nerve paralysis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2024-11-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference in discordant pairs of keratometry quality warnings between the first and third measurement | Baseline measurement (time: 0 minutes) to third study measurement (time: approximately after 6 minutes - after 3 minutes of eyelid closure) at the same study day
  As the outcome is binary (successful measurement vs. measurement with a warning/failed), the difference in discordant pairs of keratometry quality warnings between the first and third measurement

CONTACTS AND LOCATIONS:
Locations (1):
- Vienna Institute for Research in Ocular Surgery (VIROS), Department of Ophthalmology, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided
The data that support the findings of this study are available after study completion from the corresponding author upon reasonable request.